CLINICAL TRIAL: NCT00603967
Title: Aromatase Inhibitors: Skeletal Effects and the Role of CYP19 Gene Polymorphisms
Brief Title: Effect of Aromatase Inhibitors on Bones and Genes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-0918; Grant
Record Dates: First submitted 2008-01-04; First posted 2008-01-29 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Postmenopausal
Keywords: Breast Cancer; Postmenopausal; Aromatase
MeSH Terms: conditions — Breast Neoplasms | interventions — Absorptiometry, Photon; Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aromatase inhibitor (Other)
  Interventions: Procedure: Dual x-ray absorptiometry (DXA); Procedure: Blood draw; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Dual x-ray absorptiometry (DXA) — Baseline, 6 months, and 12 months
Procedure: Blood draw — Baseline - genotyping Baseline, 6 months, and 12 months - markers of bone turnover and hormonal assays
Behavioral: Questionnaire — Menopausal symptom questionnaire - baseline, 3 months, 6 months, 12 months
  Cognitive tests - baseline, 6 months, 12 months
  Depression assessment - baseline, 6 months, 12 months
  Dietary calcium intake questionnaire - baseline

SUMMARY:
The primary objective of this 2-year pilot project is to test the hypothesis that skeletal response to aromatase inhibitors is determined by polymorphisms of the CYP19 gene.

DETAILED DESCRIPTION:
A family history of osteoporosis will be noted. Data on the factors that affect estrogen exposure such as age at menarche, average number of periods per year during the reproductive years, number of years of birth control pill use, total number of pregnancies, number of pregnancies to term, months of lactation and age at menopause will be recorded. These data will be collected at baseline. Current medications and other medical problems will be recorded at baseline and during follow-up visits. New medical problems and new medications will be noted on follow-up.

Physical examination will be done at baseline and during follow-up visits. Body mass index calculated as weight (kg) divided by the square of the height (m2) will be obtained every visit. Height will be obtained using a standard stadiometer and weight will be taken using a standard weighing scale.

Dietary calcium and Vitamin D intake will be estimated from a 7-day dietary recall at baseline and adjusted to a daily intake of 1200-1500 mg of calcium per day. Vitamin D intake will also be adjusted to 800 IU per day.

Biochemical Analysis. Routine serum comprehensive metabolic profile (CMP) will be measured by standard autoanalyzer technique, serum 25-hydoxyvitamin D by double-antibody radioimmunoassay (Incstar Corp., Stillwater, Minnesota), and FSH by chemiluminescent assay (Bayer, NY) in those cases when the last menstrual period occurred less than 12 months before the signing of the informed consent. These measurements will be done through the Barnes-Jewish Hospital Laboratory. Serum estradiol will be measured by radioimmunoassay (Diagnostic Systems Laboratories Inc.), and sex hormone binding globulin by double antibody radioimmunoassay (Diagnostic Laboratories Inc). Serum estradiol measurements will be done at the Core Laboratory of the General Clinical Research Center (GCRC) of Washington University School of Medicine while the sex hormone binding globulin assay will be done at Dr. Villareal's laboratory. The inter- and intra-assay coefficients of variation for these assays are all < 10%. In order to improve accuracy of the analysis the biochemical tests (except for 25-OH Vitamin D) will be performed at the end of the study and will be run by the same operator and plate (run in batch).

Bone Mineral Density (BMD) BMD of the total body, lumbar spine and the proximal left femur will be measured by dual energy X-ray absorptiometry (DEXA) using Hologic QDR 4500 (Hologic Inc., Waltham Ma, U.S.A.). Measurements will be done at month 0, 6 and 12 (see Visits and Testing Schedule). To guarantee the necessary flexibility for the patients who can not be seen at the exact date for the follow up a window of 1 month earlier and 2 months of late will be considered. BMD of the lumbar spine will be measured from L1 to L4. The non-dominant hip will be used for studies on the proximal femur. The main regions of interest on the proximal femur will be the total femur, femoral neck and femoral trochanter. The coefficient of variability for these repeated measurements in our institution is1.09% for the lumbar spine and 1.2% for the total femur in our center.

Bone Turnover Markers will be obtained at month 0, 6 and 12. We will follow a marker of bone resorption (urine cross-linked N- telopeptide of type I collagen [urine NTx] or, when a proper 24 hour urine collection is not done, serum cross-linked telopeptide of type I collagen [serum CTx) will be analyzed) and one marker of bone formation (serum bone specific alkaline phosphatase {BSAP). Due to the diurnal pattern of bone markers, all serum specimens will be collected in the fasting state while urinary NTx will measured on 24-hour urine collection. These markers will be measured by ELISA at the Core laboratory for Clinical Studies at Washington University as follows: Urine NTX (Osteomark, Ostex International, Inc., Seattle, WA), serum CTX (serum crosslaps, Osteometer, Hawthorne, CA) and serum BSAP (Alkphase-B, Metra Biosystems, Inc., Mountain View, CA). Intra-assay coefficients of variations are in the range of 4-7% (32;33). In order to improve accuracy of the analysis biochemical tests will be performed at the end of the study and will be run by the same operator and plate (conducted in batch).

Vertebral Fracture Evaluation. We will evaluate vertebral fractures using the vertebral fracture assessment (VFA) method performed by the same DEXA machine used to measure the bone mineral density. Those patients whose VFA is suspicious for a fracture will undergo a lateral spine X-ray. Vertebral fractures will be identified by visual inspection of lateral spine radiographs of the thoracic and lumbar vertebrae, from T4 to L5. Interpretation of radiographs will be done by the PI, who is an endocrinologist specializing in bone disease and the Medical Director of the Bone Health Program in the Division of Bone and Mineral Diseases at Washington University School of Medicine. If the PI will have some doubts, she can easily ask the opinion from the bone radiologists at the Department of Radiology at Washington University School of Medicine.

Menopausal symptom evaluation. Symptoms related to menopause will be evaluated using a modified Leuven menopause questionnaire. This is a straightforward menopause-specific questionnaire which covers vasomotor, gynecologic, psychological, cognitive and somatic symptoms which was developed and validated in a previous study (Anti-Cancer Drugs 2004 15:753-760). The Leuven questionnaire includes definitions of each menopausal symptoms and rated as: 1 (no symptom), 2 (mild) up to 5 (intolerable). This questionnaire will be administered at month 0, 3, 6 and 12. This questionnaire will be administered during the patient visits at month 0, 6 and 12, and it will be sent by mail approximately two weeks prior to month 3. A phone call will also be made to the patients to prompt them to complete the questionnaire approximately at the time they should receive it by mail (month 3). Those who will fail to send the questionnaire within 1 week after the indicated dates will be contacted by phone. A log will be kept to document phone call attempts and dates of mailings to document persistence with compliance. A symptom score will be estimated for each participant. The number of symptomatic subject in each genotype will also be estimated.

Psychometric testing: In the current project we will assess the cognitive impairment using the mini mental state examination test (normal range of > 72 for women < 8 years of formal education and > 76 for those who have > 9 years of formal education) and attention and executive functions using Trail making tests A and B (the score is the number of seconds spent in connecting 25 numbered circles in sequential order [trail A] or the seconds spent in connecting numbered circles (1-13) alternately to letters of the alphabet (A-L) in sequential order [Trail B]. In both tests a maximum of 180 seconds is allowed). A fluency test will be performed asking to the subjects to name as many animals as they can during 1 minute. Additionally the Geriatric Depression Scale (GDS) will be performed in order to exclude and to assess eventual depression. This test implies 30 questions, each one corresponding to a score of 0 or 1. According to the final score a patient is classified normal with a score ranging from 0 to 9, mildly depressed if from 10 to 20, and severely depressed if the score is higher than 20. These tests will be administered during the patient visits at month 0, 6 and 12.

Rationale. To date, 4 polymorphisms of the aromatase gene have been associated with significant differences in BMD and fracture risk (16-18), age-related bone loss (18;29) a few of which have also been found to be associated with differences in breast cancer risk (30). Functional in-vitro analysis suggests an altered enzymatic activity in certain variants for this gene perhaps accounting for differences in the risk of breast cancer and osteoporosis. Variants with increased aromatase activity (18), as in those with higher number of TTTA repeats, have higher BMD but higher risk for breast cancer (30) possibly a consequence of higher estrogen levels. Because these variants have increased enzyme activity, it is possible that this select group of women will have increased sensitivity to aromatase inhibition and would experienced more bone loss than those with lower aromatase activity. On the contrary, it is also possible that women with these variant alleles will be relatively resistant to aromatase inhibition compared to variants with lower enzymatic activity and will continue to synthesize estrogen from precursors and, therefore, will not develop rapid bone loss. This proposal will address this important question by comparing the variants of the different polymorphisms described below.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged greater than or equal to 40 years, at least 12 months from last menstrual period. For subjects who are amenorrheic for < 12 months (including patients who had hysterectomy, received ERT/HRT, or rendered amenorrheic by chemotherapy), they must have serum FSH =50 UI/L.
* Must have diagnosis of breast cancer stages I-IIIA.
* Planned therapy for the treatment group must include aromatase inhibitors using third generation non-steroidal aromatase inhibitors, anastrozole or letrozole. Those who are already treated with aromatase inhibitors and have bone density measurements prior to initiation of aromatase inhibitors or will be switched from tamoxifen to third generation aromatase inhibitors will also be included in the study.
* Bone mineral density measurement must range from normal to osteopenia (T-scores between +2.0/-2.0). Those with T-scores of <-2.0 in either the lumbar spine or the femoral neck as well as those with a history of osteoporosis-related fractures or vertebral deformities on lateral spine radiographs will be excluded from the study.
* Must be ambulatory willing and able to provide informed consent.

Exclusion Criteria:

* No current use of medications affecting bone metabolism, namely: estrogen, raloxifene, tamoxifen, bisphosphonates, GnRH analogues, glucocorticoids of at least 5 mg daily for 1 month or more, anabolic steroids and dilantin.
* No evidence of diseases known to interfere with bone metabolism, such as hyperparathyroidism, hyperthyroidism, osteomalacia, chronic liver disease, renal failure, hypercortisolism, malabsorption, and immobilization.
* No current alcohol or tobacco abuse.
* No evidence of bone metastasis or evidence of abnormal clinical laboratory parameters that are assessed as clinically significant by the investigator.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Skeletal effects of aromatase inhibitors in postmenopausal women with estrogen receptor positive breast cancer. | 2 years
Influence of polymorphisms of the CYP19 gene on the skeletal response to aromatase inhibitors. | 2 years

SECONDARY OUTCOMES:
Influence of the CYP19 gene polymorphisms on the menopausal symptoms in women on aromatase inhibitor therapy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Rastelli, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Campos SM. Aromatase inhibitors for breast cancer in postmenopausal women. Oncologist. 2004;9(2):126-36. doi: 10.1634/theoncologist.9-2-126. PMID 15047917
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Baum M, Budzar AU, Cuzick J, Forbes J, Houghton JH, Klijn JG, Sahmoud T; ATAC Trialists' Group. Anastrozole alone or in combination with tamoxifen versus tamoxifen alone for adjuvant treatment of postmenopausal women with early breast cancer: first results of the ATAC randomised trial. Lancet. 2002 Jun 22;359(9324):2131-9. doi: 10.1016/s0140-6736(02)09088-8. PMID 12090977
- [Background] Howell A, Cuzick J, Baum M, Buzdar A, Dowsett M, Forbes JF, Hoctin-Boes G, Houghton J, Locker GY, Tobias JS; ATAC Trialists' Group. Results of the ATAC (Arimidex, Tamoxifen, Alone or in Combination) trial after completion of 5 years' adjuvant treatment for breast cancer. Lancet. 2005 Jan 1-7;365(9453):60-2. doi: 10.1016/S0140-6736(04)17666-6. PMID 15639680
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341
- [Background] Coombes RC, Hall E, Gibson LJ, Paridaens R, Jassem J, Delozier T, Jones SE, Alvarez I, Bertelli G, Ortmann O, Coates AS, Bajetta E, Dodwell D, Coleman RE, Fallowfield LJ, Mickiewicz E, Andersen J, Lonning PE, Cocconi G, Stewart A, Stuart N, Snowdon CF, Carpentieri M, Massimini G, Bliss JM, van de Velde C; Intergroup Exemestane Study. A randomized trial of exemestane after two to three years of tamoxifen therapy in postmenopausal women with primary breast cancer. N Engl J Med. 2004 Mar 11;350(11):1081-92. doi: 10.1056/NEJMoa040331. PMID 15014181
- [Background] Bonneterre J, Thurlimann B, Robertson JF, Krzakowski M, Mauriac L, Koralewski P, Vergote I, Webster A, Steinberg M, von Euler M. Anastrozole versus tamoxifen as first-line therapy for advanced breast cancer in 668 postmenopausal women: results of the Tamoxifen or Arimidex Randomized Group Efficacy and Tolerability study. J Clin Oncol. 2000 Nov 15;18(22):3748-57. doi: 10.1200/JCO.2000.18.22.3748. PMID 11078487
- [Background] Vergote I, Bonneterre J, Thurlimann B, Robertson J, Krzakowski M, Mauriac L, Koralewski L, Webster A, Steinberg M, von Euler M. Randomised study of anastrozole versus tamoxifen as first-line therapy for advanced breast cancer in postmenopausal women. Eur J Cancer. 2000 Sep;36 Suppl 4:S84-5. doi: 10.1016/s0959-8049(00)00239-2. PMID 11056332
- [Background] Mouridsen H, Sun Y, Gershanovich M, Perez-Carrion R, Becquart D, Chaudri-Ross HA, Lang R. Superiority of letrozole to tamoxifen in the first-line treatment of advanced breast cancer: evidence from metastatic subgroups and a test of functional ability. Oncologist. 2004;9(5):489-96. doi: 10.1634/theoncologist.9-5-489. PMID 15477633
- [Background] Paridaens R, Dirix L, Lohrisch C, Beex L, Nooij M, Cameron D, Biganzoli L, Cufer T, Duchateau L, Hamilton A, Lobelle JP, Piccart M; European Organization for the Research and Treatment of Cancer (EORTC)- Investigational Drug Branch for Breast Cancer (IDBBC). Mature results of a randomized phase II multicenter study of exemestane versus tamoxifen as first-line hormone therapy for postmenopausal women with metastatic breast cancer. Ann Oncol. 2003 Sep;14(9):1391-8. doi: 10.1093/annonc/mdg362. PMID 12954578
- [Background] Forney JP, Milewich L, Chen GT, Garlock JL, Schwarz BE, Edman CD, MacDonald PC. Aromatization of androstenedione to estrone by human adipose tissue in vitro. Correlation with adipose tissue mass, age, and endometrial neoplasia. J Clin Endocrinol Metab. 1981 Jul;53(1):192-9. doi: 10.1210/jcem-53-1-192. No abstract available. PMID 7240376
- [Background] Heshmati HM, Khosla S, Robins SP, O'Fallon WM, Melton LJ 3rd, Riggs BL. Role of low levels of endogenous estrogen in regulation of bone resorption in late postmenopausal women. J Bone Miner Res. 2002 Jan;17(1):172-8. doi: 10.1359/jbmr.2002.17.1.172. PMID 11771665
- [Background] Leelawattana R, Ziambaras K, Roodman-Weiss J, Lyss C, Wagner D, Klug T, Armamento-Villareal R, Civitelli R. The oxidative metabolism of estradiol conditions postmenopausal bone density and bone loss. J Bone Miner Res. 2000 Dec;15(12):2513-20. doi: 10.1359/jbmr.2000.15.12.2513. PMID 11127217
- [Background] Masi L, Becherini L, Gennari L, Amedei A, Colli E, Falchetti A, Farci M, Silvestri S, Gonnelli S, Brandi ML. Polymorphism of the aromatase gene in postmenopausal Italian women: distribution and correlation with bone mass and fracture risk. J Clin Endocrinol Metab. 2001 May;86(5):2263-9. doi: 10.1210/jcem.86.5.7450. PMID 11344237
- [Background] Somner J, McLellan S, Cheung J, Mak YT, Frost ML, Knapp KM, Wierzbicki AS, Wheeler M, Fogelman I, Ralston SH, Hampson GN. Polymorphisms in the P450 c17 (17-hydroxylase/17,20-Lyase) and P450 c19 (aromatase) genes: association with serum sex steroid concentrations and bone mineral density in postmenopausal women. J Clin Endocrinol Metab. 2004 Jan;89(1):344-51. doi: 10.1210/jc.2003-030164. PMID 14715870
- [Background] Gennari L, Masi L, Merlotti D, Picariello L, Falchetti A, Tanini A, Mavilia C, Del Monte F, Gonnelli S, Lucani B, Gennari C, Brandi ML. A polymorphic CYP19 TTTA repeat influences aromatase activity and estrogen levels in elderly men: effects on bone metabolism. J Clin Endocrinol Metab. 2004 Jun;89(6):2803-10. doi: 10.1210/jc.2003-031342. PMID 15181061
- [Background] Tofteng CL, Kindmark A, Brandstrom H, Abrahamsen B, Petersen S, Stiger F, Stilgren LS, Jensen JE, Vestergaard P, Langdahl BL, Mosekilde L; Danish Osteoporosis Prevention Study. Polymorphisms in the CYP19 and AR genes--relation to bone mass and longitudinal bone changes in postmenopausal women with or without hormone replacement therapy: The Danish Osteoporosis Prevention Study. Calcif Tissue Int. 2004 Jan;74(1):25-34. doi: 10.1007/s00223-002-2158-3. Epub 2003 Oct 2. PMID 14517714
- [Background] Ravdin PM, Green S, Dorr TM, McGuire WL, Fabian C, Pugh RP, Carter RD, Rivkin SE, Borst JR, Belt RJ, et al. Prognostic significance of progesterone receptor levels in estrogen receptor-positive patients with metastatic breast cancer treated with tamoxifen: results of a prospective Southwest Oncology Group study. J Clin Oncol. 1992 Aug;10(8):1284-91. doi: 10.1200/JCO.1992.10.8.1284. PMID 1634918
- [Background] Tamoxifen for early breast cancer: an overview of the randomised trials. Early Breast Cancer Trialists' Collaborative Group. Lancet. 1998 May 16;351(9114):1451-67. PMID 9605801
- [Background] Osborne CK. Tamoxifen in the treatment of breast cancer. N Engl J Med. 1998 Nov 26;339(22):1609-18. doi: 10.1056/NEJM199811263392207. No abstract available. PMID 9828250
- [Background] Nabholtz JM, Buzdar A, Pollak M, Harwin W, Burton G, Mangalik A, Steinberg M, Webster A, von Euler M. Anastrozole is superior to tamoxifen as first-line therapy for advanced breast cancer in postmenopausal women: results of a North American multicenter randomized trial. Arimidex Study Group. J Clin Oncol. 2000 Nov 15;18(22):3758-67. doi: 10.1200/JCO.2000.18.22.3758. PMID 11078488
- [Background] Webb PM, Cummings MC, Bain CJ, Furnival CM. Changes in survival after breast cancer: improvements in diagnosis or treatment? Breast. 2004 Feb;13(1):7-14. doi: 10.1016/S0960-9776(03)00129-2. PMID 14759710
- [Background] Goss PE, Qi S, Josse RG, Pritzker KP, Mendes M, Hu H, Waldman SD, Grynpas MD. The steroidal aromatase inhibitor exemestane prevents bone loss in ovariectomized rats. Bone. 2004 Mar;34(3):384-92. doi: 10.1016/j.bone.2003.11.006. PMID 15003786
- [Background] Zarrabeitia MT, Hernandez JL, Valero C, Zarrabeitia AL, Garcia-Unzueta M, Amado JA, Gonzalez-Macias J, Riancho JA. A common polymorphism in the 5'-untranslated region of the aromatase gene influences bone mass and fracture risk. Eur J Endocrinol. 2004 May;150(5):699-704. doi: 10.1530/eje.0.1500699. PMID 15132727
- [Background] Kristensen VN, Harada N, Yoshimura N, Haraldsen E, Lonning PE, Erikstein B, Karesen R, Kristensen T, Borresen-Dale AL. Genetic variants of CYP19 (aromatase) and breast cancer risk. Oncogene. 2000 Mar 2;19(10):1329-33. doi: 10.1038/sj.onc.1203425. PMID 10713674
- [Background] Van Pottelbergh I, Goemaere S, Kaufman JM. Bioavailable estradiol and an aromatase gene polymorphism are determinants of bone mineral density changes in men over 70 years of age. J Clin Endocrinol Metab. 2003 Jul;88(7):3075-81. doi: 10.1210/jc.2002-021691. PMID 12843146
- [Background] Kristensen VN, Andersen TI, Lindblom A, Erikstein B, Magnus P, Borresen-Dale AL. A rare CYP19 (aromatase) variant may increase the risk of breast cancer. Pharmacogenetics. 1998 Feb;8(1):43-8. doi: 10.1097/00008571-199802000-00006. PMID 9511180
- [Background] Grodin JM, Siiteri PK, MacDonald PC. Source of estrogen production in postmenopausal women. J Clin Endocrinol Metab. 1973 Feb;36(2):207-14. doi: 10.1210/jcem-36-2-207. No abstract available. PMID 4688315
- [Background] Armamento-Villareal RC, Napoli N, Klug T, Civitelli R. The oxidative metabolism of estrogen modulates response to ERT/HRT in postmenopausal women. Bone. 2004 Sep;35(3):682-8. doi: 10.1016/j.bone.2004.05.010. PMID 15336604
- [Background] Martucci CP, Fishman J. P450 enzymes of estrogen metabolism. Pharmacol Ther. 1993 Feb-Mar;57(2-3):237-57. doi: 10.1016/0163-7258(93)90057-k. PMID 8361994
- [Background] Badawi AF, Cavalieri EL, Rogan EG. Role of human cytochrome P450 1A1, 1A2, 1B1, and 3A4 in the 2-, 4-, and 16alpha-hydroxylation of 17beta-estradiol. Metabolism. 2001 Sep;50(9):1001-3. doi: 10.1053/meta.2001.25592. PMID 11555828
- [Background] Napoli N, Villareal DT, Mumm S, Halstead L, Sheikh S, Cagaanan M, Rini GB, Armamento-Villareal R. Effect of CYP1A1 gene polymorphisms on estrogen metabolism and bone density. J Bone Miner Res. 2005 Feb;20(2):232-9. doi: 10.1359/JBMR.041110. Epub 2004 Nov 16. PMID 15647817
- [Background] Goss PE, Qi S, Cheung AM, Hu H, Mendes M, Pritzker KP. Effects of the steroidal aromatase inhibitor exemestane and the nonsteroidal aromatase inhibitor letrozole on bone and lipid metabolism in ovariectomized rats. Clin Cancer Res. 2004 Sep 1;10(17):5717-23. doi: 10.1158/1078-0432.CCR-04-0438. PMID 15355898
- [Background] Vanderschueren D, Boonen S, Ederveen AG, de Coster R, Van Herck E, Moermans K, Vandenput L, Verstuyf A, Bouillon R. Skeletal effects of estrogen deficiency as induced by an aromatase inhibitor in an aged male rat model. Bone. 2000 Nov;27(5):611-7. doi: 10.1016/s8756-3282(00)00363-x. PMID 11062346
- [Background] Kanis JA. Diagnosis of osteoporosis and assessment of fracture risk. Lancet. 2002 Jun 1;359(9321):1929-36. doi: 10.1016/S0140-6736(02)08761-5. PMID 12057569
- [Background] Villareal DT, Binder EF, Williams DB, Schechtman KB, Yarasheski KE, Kohrt WM. Bone mineral density response to estrogen replacement in frail elderly women: a randomized controlled trial. JAMA. 2001 Aug 15;286(7):815-20. doi: 10.1001/jama.286.7.815. PMID 11497535
- [Background] Villareal DT, Holloszy JO, Kohrt WM. Effects of DHEA replacement on bone mineral density and body composition in elderly women and men. Clin Endocrinol (Oxf). 2000 Nov;53(5):561-8. doi: 10.1046/j.1365-2265.2000.01131.x. PMID 11106916
- [Background] Guthrie JR, Ebeling PR, Hopper JL, Barrett-Connor E, Dennerstein L, Dudley EC, Burger HG, Wark JD. A prospective study of bone loss in menopausal Australian-born women. Osteoporos Int. 1998;8(3):282-90. doi: 10.1007/s001980050066. PMID 9797914
- [Background] Armamento-Villareal R, Civitelli R. Estrogen action on the bone mass of postmenopausal women is dependent on body mass and initial bone density. J Clin Endocrinol Metab. 1995 Mar;80(3):776-82. doi: 10.1210/jcem.80.3.7883830.
- [Background] Kado DM, Browner WS, Blackwell T, Gore R, Cummings SR. Rate of bone loss is associated with mortality in older women: a prospective study. J Bone Miner Res. 2000 Oct;15(10):1974-80. doi: 10.1359/jbmr.2000.15.10.1974. PMID 11028450